CLINICAL TRIAL: NCT00252668
Title: An Open-Label, Multicentre, Extension Study of the Combination of Etanercept and Methotrexate in Rheumatoid Arthritis Subjects
Brief Title: Study Evaluating the Combination of Etanercept and Methotrexate in Rheumatoid Arthritis Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0881A1-101631; B1801221; 0881A1-400
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2011-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept; Methotrexate

INTERVENTIONS:
Drug: Etanercept
Drug: Methotrexate

SUMMARY:
This study is an open label extension of a previously completed double-blind, randomized study comparing etanercept and methotrexate in subjects with active rheumatoid arthritis. All subjects will receive combination treatment with etanercept and methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who completed the previous double-blind,randomized study.
* Ability to reconstitute and self-inject test etanercept (ETN) or have a designee who can do so.

Exclusion Criteria:

* Dose of prednisone>10 mg/day (or equivalent) or dose changed within 2 weeks before week 0 evaluation.
* Clinically relevant concurrent medical events including: uncompensated congestive heart failure (CHF), diagnosis of multiple sclerosis or other central demyelinating diseases, presence or history of confirmed blood dyscrasias, cancer or history of cancer, serious infection within 1 month of test article administration or active infection at week 0.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-06; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the long-term safety of the combination of etanercept and methotrexate in adults with RA who have completed the previous double-blind, randomized study.

SECONDARY OUTCOMES:
To evaluate the long-term clinical efficacy and x-ray progression of the combination of etanercept and methotrexate in adults with RA who have completed the previous double-blind, randomized study.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Germany, MedinfoDEU@wyeth.com; Trial Manager, Principal Investigator — For Sweden, Denmark and Norway, MedInfoNord@wyeth.com; Trial Manager, Principal Investigator — For Belgium, trials-BEL@wyeth.com; Trial Manager, Principal Investigator — For Greece, decresg@wyeth.com; Trial Manager, Principal Investigator — For Czech Republic, WPPGCLI@wyeth.com; Trial Manager, Principal Investigator — For Romania, WPVIMED@wyeth.com; Trial Manager, Principal Investigator — For Poland, WPWZMED@wyeth.com; Trial Manager, Principal Investigator — For Spain, Italy, Portugal, the Netherlands, and Finland, clinicaltrialinfo@wyeth.com